CLINICAL TRIAL: NCT04617431
Title: Application of Wearable Devices to Build a Self-Management Model in Chronic Kidney Disease Patients- Analysis of Healthcare Cost
Brief Title: Application of Wearable Devices to Build a Self-Management Model in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201808094RINB
Record Dates: First submitted 2020-06-07; First posted 2020-11-05 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention involved reminding the intervention group to upload their dietary diary every day. The researchers were trained by a dietitian and provided suggestions about diet and exercise to the intervention group. "LINE " is a mobile app operated by LINE Corporation. All users can use texts, images, video, and audio for contact at any time. A LINE group was created to deliver medical knowledge of diet and exercise. Each of the messages were guided by a diet manual for kidney disease (edited by Department of Dietetics, National Taiwan University Hospital Yunlin Branch). The intervention group also asked questions about CKD management, and a teleconsultation of health information was provided. A daily target of 7,500 steps was set and used to emphasize the correct concepts about exercise. Participants were inspired in the intervention group if someone achieved the target number of steps.
  Interventions: Behavioral: Mobile health application and social media
- Control group (No Intervention): The participants of control group had a wearable device and could upload their dietary diary to the health management platform every day. But no "LINE" group was created, and no reminding.

INTERVENTIONS:
Behavioral: Mobile health application and social media — The intervention involved reminding the intervention group to upload their dietary diary every day. The researchers were trained by a dietitian and provided suggestions about diet and exercise to the intervention group. "LINE " is a mobile app operated by LINE Corporation. All users can use texts, images, video, and audio for contact at any time. A LINE group was created to deliver medical knowledge of diet and exercise. Each of the messages were guided by a diet manual for kidney disease (edited by Department of Dietetics, National Taiwan University Hospital Yunlin Branch). The intervention group also asked questions about CKD management, and a teleconsultation of health information was provided. A daily target of 7,500 steps was set and used to emphasize the correct concepts about exercise. Participants were inspired in the intervention group if someone achieved the target number of steps.
  Arms: Intervention group

SUMMARY:
Aim: By application of wearable devices and health management platform to build self-management model in CKD patients and analyze the cost of healthcare.

Material and Methods: The investigators plan to recruit 60 CKD patients as trial subjects. The intervention group is composed of 30 participants, and the control group 30 participants. The intervention group received intervention with wearable devices and health management platform for 90 days. Patients record diet diary by a smartphone application, and their exercise-related data are collected by wearable devices. Then, all the collected information will be upload to health management platform. The investigators also create a LINE group to encourage exercise in the experimental group. The investigators compare the scores of self-management sheet and physical and laboratory examinations before and after the intervention. The investigators also analyze the cost of healthcare within 180 days.

DETAILED DESCRIPTION:
Background: End stage renal disease (ESRD) is a global public health issue. The dialysis therapy brings huge economic burden to many countries. According to the report of 2015 United States Renal Data System (USRDS), the incidence rate of ESRD is 458 people per million populations. And the prevalence rate is 3,138 people per million populations, which is the highest one in the world. Chronic kidney disease (CKD) can be classified into five stages according to glomerular filtration rate. Whatever the stage it is, patients should keep healthy habits about diet and exercise and good adherence to medication. If patients are able to monitor their lifestyle, it not only promotes health, but also reduces the cost of health care.

Aim: By application of wearable devices and health management platform to build self-management model in CKD patients and analyze the cost of healthcare.

Material and Methods: The investigators plan to recruit 60 CKD patients as trial subjects. The intervention group is composed of 30 participants, and the control group 30 participants. The intervention group received intervention with wearable devices and health management platform for 90 days. Patients record their own diet diary by a smartphone application, and their exercise-related data are collected by wearable devices. Then, all the collected information will be upload to health management platform. The investigators also create a LINE group to encourage exercise in the experimental group. The investigators compare the scores of self-management sheet and physical and laboratory examinations before and after the intervention. The investigators also analyze the cost of healthcare within 180 days.

ELIGIBILITY:
Inclusion Criteria

* Chronic kidney disease stage 1-4
* Agree to partake in the study signed informed consent forms for participation.

Exclusion Criteria:

* Can not use a smartphone
* Have impaired walking capacity
* Psychiatric disorder
* Have been hospitalized during the previous three months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Self-efficacy at 3 months | (1) baseline, (2) after the 90-day intervention
  the score of self-efficacy questionnaire (score 0-200, the higher the better) in units
Change from Baseline Self-management at 3 months | (1) baseline, (2) after the 90-day intervention
  the score of self-management questionnaire (score 16-64, the higher the better) in units
Change from Baseline Quality of life score at 3 months | (1) baseline, (2) after the 90-day intervention
  the score of Kidney Disease Quality of Life (KDQOL-SF™) questionnaire (score 74-360, the higher the better) in units
Change from Baseline Body composition at 3 month | (1) baseline, (2) after the 90-day intervention
  weight and height will be combined to report BMI in kg/m^2
Change from Baseline Renal function at 3 months | (1) baseline, (2) after the 90-day intervention
  estimated glomerular filtration rate in mL/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yi Li, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li WY, Chiu FC, Zeng JK, Li YW, Huang SH, Yeh HC, Cheng BW, Yang FJ. Mobile Health App With Social Media to Support Self-Management for Patients With Chronic Kidney Disease: Prospective Randomized Controlled Study. J Med Internet Res. 2020 Dec 15;22(12):e19452. doi: 10.2196/19452. PMID 33320101